CLINICAL TRIAL: NCT05626283
Title: Transforaminal Epidural Steroid Injection in Lumbar Disc Prolapse: Impact on Pain and Cognition in Relation to Micro RNA-155 Serum Level
Brief Title: Impact of Transforaminal Epidural Steroid Injection in Lumbar Disc Prolpse on Micro RNA-155 Serum Level
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mona Hussein, Associate professor of Neurology, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/050722022/Mohiee
Record Dates: First submitted 2022-11-04; First posted 2022-11-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lumbar disc prolapse group (Active Comparator): 44 patients diagnosed as having symptomatic lumbar disc prolapse
  Interventions: Drug: transforaminal epidural injection.; Other: micro RNA-155 serum level
- Control (Placebo Comparator): 44 age and sex matched healthy controls
  Interventions: Other: micro RNA-155 serum level

INTERVENTIONS:
Drug: transforaminal epidural injection. — transforaminal epidural steroid injection.
  Arms: lumbar disc prolapse group
Other: micro RNA-155 serum level — Estimation of miR-155 expression level:

SUMMARY:
Chronic pain could be considered a brain disease as it can affect multiple aspects of brain function, chemistry, neural networks and structure. Pain is associated with impaired cognitive function (1). Around 45-50% of these patients report cognitive deficits such as forgetfulness (23.4%), minor accidents (23.1%), difficulty finishing tasks (20.5%), and difficulty maintaining attention (18.7%) (2,3). Many studies emphasised an impairment in the cognitive tests assessing executive functioning, attention abilities, processing speed, and memory in patients with chronic pain (4,5). Studies of community-dwelling older adults found that pain, particularly widespread or severe pain, was associated with mobility Limitations in physical performance (e.g., walking speed, stair climbing, and activities of daily living) (6-9) in individuals with chronic pain and correspond to the pain level (10,11). Finally, both pain and impaired cognition affect mobility status in older adults, and mobility is affected to a greater extent when both are present (12).

Recent data indicate that miR-155 has a typical multifunctional miRNA and plays a crucial role in various physiological and pathological processes such as immunity, inflammation, cognitive dysfunction and neuropathies (13). The available experimental evidence indicating that miR-155 is up-regulated in neuropathies allows us to include this miRNA in the list of genes of paramount importance in chronic low back pain diagnosis and prognosis. Exogenous molecular control in vivo of miR-155 expression could open up new ways to restore cognitive outcome or attenuate the pain intensity (14).

No study searched the role of intervention (epidural steroid injection) on cognitive function reserve, whether it is a better substitution or not for the conservative medical treatment. Since exogenous steroid is a part of epidural injection, the systemic effect of a single dose of steroids does not affect cognitive function, giving superiority to the intervention modality on the conservative medical therapy approach (15).

Aim ot the work This work aims to study the impact of transforaminal epidural steroid injection in lumbar disc prolapse on pain intensity and cognitive function in relation to Micro RNA-155 serum level.

DETAILED DESCRIPTION:
Study design and Participants:

The study will be conducted in two stages:

Stage (1): It will be a case control study that will include 44 patients diagnosed as having symptomatic lumbar disc prolapse and 44 age and sex matched healthy controls. Both patients and control groups will be subjected to measurement of baseline miR-155 expression level.

Stage (2): It will be an interventional non-experimental study that will include only the 44 patients who had symptomatic lumbar disc prolapse. Those patients will be subjected to transforaminal epidural steroid injection. Assessment of pain intensity, functional disability, cognitive function, depression, and miR-155 expression level will be done for the included patients before and 1 month after transforaminal epidural steroid injection to clarify the effect steroid injection on these variables.

The included patients will be recruited from the neurology and pain clinics of Beni-Suef University Hospital, in the period from December 2022 to September 2023.

The study will include patients with clinical evidence of disc bulge in the form of disc related radicular pain of >3 months duration, not responding to conservative treatment and interfering with daily activities. The selected patients should have radiological evidence of posterolateral lumbar disc bulge by MRI lumbosacral.

Data collection History will be taken from the selected patients regarding the demographics and the duration of lumbar disc related radicular pain. The imaging findings regarding the number of prolapsed discs and the degree of the most prolapsed disc will be also obtained.

Assessment of pain intensity and functional disability Assessment of the pain intensity and functional disability will be done before and 1 month after the interventional pain management procedure. Assessment will be done using Numeric Rating Scale (NRS) and Oswestry Disability Index (ODI).

Cognitive assessment Cognitive assessment will be done before and 1 month after the interventional pain management procedure. Assessment will be done using Paired Associate Learning test (PALT), Paced Auditory Serial Addition Test (PASAT), and Controlled Oral Word Association Test (COWAT).

Interventional pain Procedure:

The selected patients will be brought to the preparation room where reassurance will be done. Intravenous midazolam 0.2 mg/kg will be given to them, then they will be placed in the prone position on fluoroscopy table and draped in a sterile manner. They will be connected to a monitor (SPO2, NIBLP, and ECG) and given supplemental oxygen through a nasal cannula (3 L/min) to maintain the oxygen saturation. A 22-gauge, 3.5-inch spinal needle will be used in the injection procedure. With each insertion of the spinal needle, 1 ml with 20 mg of local anesthetic lidocaine 2% will be injected intradermally.

The patients will be given transforaminal epidural injection of steroids with local anesthetic (7 mg Betamethasone preceded by a test dose of 1 milliliter 2% lidocaine).

Laboratory assessment Estimation of miR-155 expression level: Blood samples (5 mL) will be collected from the patients (before and 1 month after the interventional procedure) and controls. The samples will be centrifuged at 3000 rpm for 10 min and plasma and/ or serum will be stored at -80 C till analysis. Total RNA will be extracted. Quantitative real-time polymerase chain reaction (PCR) will be performed. miR-155 expression level will be calculated by the difference in threshold cycle method.

ELIGIBILITY:
Inclusion criteria

• Patients with clinical and radiological evidence of L4-L5 disc prolapse manifesting as radicular pain and/or low back pain unresponsive to medical treatment and physiotherapy over a period of at least three months.

Exclusion criteria

* Patients with severe lumbar disc prolapse affecting motor or sphincteric functions,
* History of spinal surgery, spinal trauma, spinal deformities, spinal neoplasm or any spinal inflammatory lesion, hip osteoarthritis or sacroiliitis.
* Patients with medical disorders known to cause cognitive impairment
* Pregnant women were excluded

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Assessment of pain intensity | 1 month
  Change in Numeric Rating Scale following transforaminal epidural steroid injection: It is an 11-point numeric scale for pain intensity evaluation, ranging from 0 to 10, where higher scores denote more intense pain.
Assessment of functional disability | 1 month
  Change in Oswestry Disability Index following transforaminal epidural steroid injection: It consists of ten questions, scored on a scale of 0-5 for each, where higher scores denote more limitations. After the summation of all these subscores, the result is multiplied by two to gain the index (ranging from 0 to 100).
Assessment of functional disability | 1 month
  Change in Functional rating index following transforaminal epidural steroid injection: The scale consists of 10 items scored on a scale of 0-4 for each, where higher scores denote more disability.
Memory assessment | 1 month
  Change in Paired Associate Learning test following transforaminal epidural steroid injection: The test was conducted on three trials. A score of 0.5 is given for each true well-matched pair, while a score of 1 is given for each true mismatched pair, with a total score ranging between 0 and 21.
Attention assessment | 1 month
  Change in Paced Auditory Serial Addition Test following transforaminal epidural steroid injection: A set of single digits is audio recorded at a rate of one every 3 seconds and then introduced to the subject. The subject was requested to add each digit to the one just heard before. The number of correct answers was summed to gain the total score (0 to 60).
Assessment of verbal fluency and executive function. | 1 month
  Change in Controlled Oral Word Association Test following transforaminal epidural steroid injection: The subject was inquired to generate words that begin with a specified letter in one minute, eliminating proper nouns.
Assessment of miR-155 expression level | 1 month
  Change in miR-155 expression level following transforaminal epidural steroid injection.

SECONDARY OUTCOMES:
The relationship between pain intensity and functional disability, cognitive function, and miRNA-155 serum level in patients with lumbar disc prolapse. | At the same time point before intervention
  The relationship between the scores of pain intensity and functional disability scales (Numeric Rating Scale, Oswestry Disability Index, and Functional Rating Index), scores of the psychometric tests (Paired Associate Learning test, Paced Auditory Serial Addition Test, Controlled Oral Word Association Test), and miRNA-155 serum level

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Hussein, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fathy W, Hussein M, Magdy R, Nasser M, Mohamed J, Sayem DM, Elmoutaz H, Mounir N, Fakhry DM, Abdelbadie M. Transforaminal Epidural Steroid Injection in Lumbar Disc Prolapse: Impact on Pain Intensity and Cognitive Function in Relation to MicroRNA-155 Serum Level. Anesthesiol Res Pract. 2025 Apr 7;2025:2201031. doi: 10.1155/anrp/2201031. eCollection 2025. PMID 40230811